CLINICAL TRIAL: NCT05819502
Title: A Prospective Clinical Trial Evaluating the "Profile HIT" (Holistic Individualized Treatment)
Brief Title: "Profile HIT" (Holistic Individualized Treatment)
Acronym: HIT-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Principal Investigator, Andreas Nikolis, Principal Investigator, Erevna Innovations Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 02-2023-HIT-PRF
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Aesthetic
Keywords: Hyaluronic acid; Fillers; Volumization; Facial Profile; Patient Assessment

STUDY DESIGN:
Intervention Model Description: This study will consist of an open-label, prospective, cohort trial design. Eighteen subjects will be recruited. Subjects will be recruited based on their primary deficit, where all subjects must have a mild or greater deficit of the midface and each of three subsets of 6 subjects will have a primary deficit/deformity of the nose, lips, and chin. All subjects will receive active treatment with hyaluronic acid at Baseline, with an optional touch at week two. There will be no placebo or no-treatment control groups. Subjects will be followed for five months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Restylane line of injectables

INTERVENTIONS:
Drug: Restylane line of injectables — Restylane fillers are manufactured by Q-Med AB, part of the Galderma Group.

SUMMARY:
The "Holistic Individualized Treatment" (HIT) approach is used to identify treatment priorities, focus areas, and appropriate products for soft tissue filler treatments.

The "Profile HIT" considers the balance between the midface, nose, lips, and chin to improve a patient's appearance. This trial will assess the effectiveness of the Profile HIT algorithm in treating patients with different profile issues (e.g. nasal deformities, volume loss, chin retrusion).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must voluntarily sign and date an informed consent, including the photography addendum allowing unrestricted use of photographs for the benefit of marketing and educational purposes, approved by an independent ethics committee, before the initiation of any screening or study-specific procedures.
* Subjects must be adult male or female, at least 18 years old.
* Subjects must be willing and able to comply with procedures required in the protocol.
* Subjects must be in good health as per the investigator's judgment based on medical history
* Female subjects that are not pregnant or breastfeeding and are not considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of the study medical device or until the end of the study, whichever is longer.

Exclusion Criteria:

* Subject with uncontrolled systemic disease.
* Subject with or have a history of any medical condition that may place the subject at increased risk following exposure to hyaluronic acid or interfere with the study evaluation, including:

  * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
  * History of facial nerve palsy
  * Infection or dermatological condition at the treatment injection sites
  * Marked facial dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or overly photodamaged skin
* Subject with a history of clinically significant medical conditions or any other reason that the investigator determines would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive the study medical intervention
* Subjects with a history of an allergic reaction or significant sensitivity to constituents of the study medical intervention (or its excipients).
* Subjects with porphyria
* Subjects with active diseases, such as inflammation, infection or tumours, in or near the intended treatment sites,
* Subjects with bleeding disorders or taking thrombolytics or anticoagulants.
* Subjects who need to take immunosuppressants.
* Subjects with tattoos, jewelry, or clothing which obscure the treatment area and cannot be removed.
* Subjects who have anticipated the need for surgery or overnight hospitalization during the study.
* Subjects with a history of surgical procedures in the face, including any lifting method (e.g., facial lift, suture lift, thread lift, brow lift, eyelid and eyebrow surgery).
* Subjects with a history of facial treatment with semi-permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* Subjects with known active COVID infection within 14 days of baseline treatment.
* Subjects that have been treated with any investigational product within 30 days before the first dose of the study medical device or are currently enrolled in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint - Global Aesthetics Improvement Scale (GAIS) | At week 8
  Frequency of subjects having at least "improved" (e.g., "improved", "much improved" or "very much improved") on the Global Aesthetics Improvement Scale (GAIS), as graded by a blinded evaluator.

CONTACTS AND LOCATIONS:
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No